CLINICAL TRIAL: NCT00383123
Title: A Phase III, Single-blind, Randomized Study to Evaluate the Immunogenicity and Safety of Fluarix® (GSK Biologicals') Compared With Fluzone® (Aventis Pasteur/Sanofi) Administered Intramuscularly in Children (6 Months and Older)
Brief Title: Study Comparing the Immune Response and Safety of Fluarix and Fluzone Influenza Vaccines in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104858
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2008-12-04 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Fluarix; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Fluarix Group (Experimental): Subjects in this group received Fluarix™ and will be further stratified by 3 age groups
  * 1:1 in 6 months to < 36 months
  * 1:1 in 3 to < 5 years
  * 3:1 in 5 to < 18 years
  Interventions: Biological: Fluarix™
- Fluzone Group (Active Comparator): Subjects in this group received Fluzone and will be further stratified by 3 age groups
  * 1:1 in 6 months to < 36 months
  * 1:1 in 3 to < 5 years
  * 3:1 in 5 to < 18 years
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluarix™ — Subjects were administered 1 or 2 doses* intramuscularly, into the non-dominant upper arm for children > 12 months of age, in the anterolateral thigh for children < 12 months.
  *Only those subjects between the age of 6 months and < 9 years, who had no history of prior influenza vaccination, received 2 doses at months 0 & 1.
  Arms: Fluarix Group
Biological: Fluzone — Subjects were administered 1 or 2 doses* intramuscularly, into the non-dominant upper arm for children > 12 months of age, in the anterolateral thigh for children < 12 months.
  *Only those subjects between the age of 6 months and < 9 years, who had no history of prior influenza vaccination, received 2 doses at months 0 & 1.
  Arms: Fluzone Group

SUMMARY:
The purpose of this study is to compare two influenza vaccines (Fluzone and Fluarix) in terms of the immune response elicited and safety with a six month follow-up after first vaccination. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child age 6 months to < 18 years at the time of the vaccination; children who may or may not have had previous administration of influenza vaccine in a previous season are acceptable.
* Subjects having a parent/guardian who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the subject's parent/guardian; assent obtained in subjects > 10 years.
* Female subjects of childbearing potential must agree to take a pregnancy test.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine, other than the study vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period. Routine, registered childhood vaccinations are not an exclusion.
* History of hypersensitivity to any vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrollment.
* History of Guillain Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Pregnant or lactating female.
* Receipt of an influenza vaccine outside of this study, during current (2006-07) flu season.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3327 (Actual)
Dates: Start 2006-11-02; Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (38):
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Fairfield, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Richmond, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Tifton, Georgia
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Fishkill, New York
  - GSK Investigational Site, Hopewell Junction, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li-Kim-Moy J, Wood N, Jones C, Macartney K, Booy R. Impact of Fever and Antipyretic Use on Influenza Vaccine Immune Reponses in Children. Pediatr Infect Dis J. 2018 Oct;37(10):971-975. doi: 10.1097/INF.0000000000001949. PMID 29465480
- [Derived] Baxter R, Jeanfreau R, Block SL, Blatter M, Pichichero M, Jain VK, Dewe W, Innis BL. A Phase III evaluation of immunogenicity and safety of two trivalent inactivated seasonal influenza vaccines in US children. Pediatr Infect Dis J. 2010 Oct;29(10):924-30. doi: 10.1097/INF.0b013e3181e075be. PMID 20431425
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects, enrolled in the Fluzone Group, were not vaccinated; therefore, they were not included in the number of subjects included under "STARTED".
Groups:
- Fluarix Group: Subjects in this group received Fluarix and will be further stratified by 3 age groups
  * 1:1 in 6 months to < 36 months
  * 1:1 in 3 to < 5 years
  * 3:1 in 5 to < 18 years
Period: Overall Study
Arm/Group | Fluarix Group | Fluzone Group
Started | 2115 | 1210
Completed | 2004 | 1124
Not Completed | 111 | 86
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 68 | 61
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 27 | 18
Not completed — Other reason | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Group | Fluzone Group | Total
Number analyzed (Participants) | 2115 | 1210 | 3325
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (4.97) | 5.5 (4.75) | 6.8 (4.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1038 | 586 | 1624
  Male | 1077 | 624 | 1701
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage / african american | 344 | 238 | 582
  American indian or alaskan native | 78 | 45 | 123
  Asian - central/south asian heritage | 13 | 7 | 20
  Asian - east asian heritage | 15 | 13 | 28
  Asian - japanese heritage | 3 | 1 | 4
  Asian - south east asian heritage | 21 | 17 | 38
  Native hawaiian or other pacific island | 14 | 10 | 24
  White - arabic / north african heritage | 29 | 17 | 46
  White - caucasian / european heritage | 1477 | 794 | 2271
  Unspecified | 121 | 68 | 189

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Serum Haemagglutination-inhibition (HI) Antibodies
Description: GMTs and their 95% confidence interval are presented for all 3 viral strains comprised in the vaccine.
Time Frame: 21 or 28 days after last vaccine dose
Population: Per protocol, GMTs were assessed only in part of the According-To-Protocol (ATP) cohort for immunogenicity (children aged 6 months to < 5 years).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 426 | 445
Titer
  A/New Caledonia [6 to <36 months]: number analyzed (Participants) | 206 | 224
  A/New Caledonia [6 to <36 months] | 52.4 [43.3 to 63.4] | 101.4 [86.9 to 118.2]
  A/Wisconsin [6 to <36 months]: number analyzed (Participants) | 206 | 224
  A/Wisconsin [6 to <36 months] | 80.5 [62.2 to 104.1] | 218.0 [185.8 to 255.8]
  B/Malaysia [6 to <36 months]: number analyzed (Participants) | 206 | 224
  B/Malaysia [6 to <36 months] | 20.2 [15.9 to 25.8] | 40.6 [32.3 to 51.1]
  A/New Caledonia [3 to < 5 years]: number analyzed (Participants) | 220 | 221
  A/New Caledonia [3 to < 5 years] | 130.3 [108.6 to 156.4] | 168.7 [138.7 to 205.2]
  A/Wisconsin [3 to < 5 years]: number analyzed (Participants) | 220 | 221
  A/Wisconsin [3 to < 5 years] | 458.1 [365.3 to 574.3] | 483.4 [396.8 to 588.9]
  B/Malaysia [3 to < 5 years]: number analyzed (Participants) | 220 | 221
  B/Malaysia [3 to < 5 years] | 54.9 [42.3 to 71.1] | 64.4 [49.5 to 83.8]

2. Primary Outcome: Number of Seroconverted Subjects
Description: Seroconverted subjects are defined as subjects with either a pre-vaccination HI titer <1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum 4-fold increase at post-vaccination titer.
  Data are presented for all 3 viral strains comprised in the vaccine.
Time Frame: 21 or 28 days after last vaccine dose
Population: As per protocol, seroconversion was assessed in part of the ATP cohort for immunogenicity: children aged 6 months to < 5 years for whom post-vaccination results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 425 | 443
Participants
  A/New Caledonia [6 to <36 months]: number analyzed (Participants) | 205 | 223
  A/New Caledonia [6 to <36 months] | 105 | 179
  A/Wisconsin [6 to <36 months]: number analyzed (Participants) | 205 | 223
  A/Wisconsin [6 to <36 months] | 117 | 190
  B/Malaysia [6 to <36 months]: number analyzed (Participants) | 205 | 223
  B/Malaysia [6 to <36 months] | 48 | 114
  A/New Caledonia [3 to <5 years]: number analyzed (Participants) | 220 | 220
  A/New Caledonia [3 to <5 years] | 160 | 159
  A/Wisconsin [3 to <5 years]: number analyzed (Participants) | 220 | 220
  A/Wisconsin [3 to <5 years] | 156 | 155
  B/Malaysia [3 to <5 years]: number analyzed (Participants) | 220 | 220
  B/Malaysia [3 to <5 years] | 117 | 122

3. Primary Outcome: Number of Subjects Reporting Rare Serious Events
Description: Rare serious event is defined as any untoward medical event with an occurrence rate of ≥1/300 that:
  * resulted in death,
  * was life-threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity, or
  * was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to 6 months after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 2115 | 1210
Participants | 11 | 11

4. Secondary Outcome: Number of Seroprotected Subjects
Description: Seroprotected subjects are defined as vaccinees with a serum HI titer ≥ 1:40. Data are presented for all 3 viral strains comprised in the vaccine.
Time Frame: Before (PRE) and 21 or 28 days after (POST) the last vaccine dose
Population: As per protocol, seroprotection was assessed in part of the ATP cohort for immunogenicity: children aged 6 months to < 5 years for whom results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 426 | 445
Participants
  A/New Caledonia [6 to <36 months] PRE: number analyzed (Participants) | 205 | 223
  A/New Caledonia [6 to <36 months] PRE | 15 | 16
  A/New Caledonia [6 to <36 months] POST: number analyzed (Participants) | 206 | 224
  A/New Caledonia [6 to <36 months] POST | 122 | 193
  A/Wisconsin [6 to <36 months] PRE: number analyzed (Participants) | 205 | 223
  A/Wisconsin [6 to <36 months] PRE | 39 | 44
  A/Wisconsin [6 to <36 months] POST: number analyzed (Participants) | 206 | 224
  A/Wisconsin [6 to <36 months] POST | 135 | 211
  B/Malaysia [6 to <36 months] PRE: number analyzed (Participants) | 205 | 223
  B/Malaysia [6 to <36 months] PRE | 11 | 12
  B/Malaysia [6 to <36 months] POST: number analyzed (Participants) | 206 | 224
  B/Malaysia [6 to <36 months] POST | 50 | 115
  A/New Caledonia [3 to <5 years] PRE: number analyzed (Participants) | 220 | 220
  A/New Caledonia [3 to <5 years] PRE | 38 | 45
  A/New Caledonia [3 to <5 years] POST: number analyzed (Participants) | 220 | 221
  A/New Caledonia [3 to <5 years] POST | 180 | 189
  A/Wisconsin [3 to <5 years] PRE: number analyzed (Participants) | 220 | 220
  A/Wisconsin [3 to <5 years] PRE | 131 | 122
  A/Wisconsin [3 to <5 years] POST: number analyzed (Participants) | 220 | 221
  A/Wisconsin [3 to <5 years] POST | 194 | 207
  B/Malaysia [3 to <5 years] PRE: number analyzed (Participants) | 220 | 220
  B/Malaysia [3 to <5 years] PRE | 30 | 26
  B/Malaysia [3 to <5 years] POST: number analyzed (Participants) | 220 | 221
  B/Malaysia [3 to <5 years] POST | 121 | 129

5. Secondary Outcome: Number of Initially Unprotected Subjects With at Least a 4 Fold Increase in HI Titer
Description: Initially unprotected subjects are subjects with a baseline HI titer < 1:40. Data are presented for all 3 viral strains comprised in the vaccine.
Time Frame: 21 or 28 days after last vaccine dose
Population: As per protocol, only subjects from the ATP cohort for immunogenicity aged 6 months to < 5 years and with a baseline titre < 1:40 were analysed for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 384 | 405
Participants
  A/New Caledonia [6 to <36 months]: number analyzed (Participants) | 190 | 207
  A/New Caledonia [6 to <36 months] | 125 | 117
  A/Wisconsin [6 to <36 months]: number analyzed (Participants) | 166 | 179
  A/Wisconsin [6 to <36 months] | 114 | 173
  B/Malaysia [6 to <36 months]: number analyzed (Participants) | 194 | 211
  B/Malaysia [6 to <36 months] | 74 | 129
  A/New Caledonia [3 to <5 years]: number analyzed (Participants) | 182 | 175
  A/New Caledonia [3 to <5 years] | 163 | 155
  A/Wisconsin [3 to <5 years]: number analyzed (Participants) | 89 | 98
  A/Wisconsin [3 to <5 years] | 75 | 92
  B/Malaysia [3 to <5 years]: number analyzed (Participants) | 190 | 194
  B/Malaysia [3 to <5 years] | 115 | 125

6. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness, and swelling. Solicited general symptoms assessed include drowsiness, fever, irritability, loss of appetite, arthralgia, fatigue, headache, muscle aches, and shivering.
  Data across doses are presented. Any = at least one symptom irrespective of intensity/relationship to vaccination; Grade 3: symptom that prevented normal everyday activities; Related: considered by the investigator as related to the study vaccination.
Time Frame: During a 4-day follow-up period after each vaccination
Population: Analysis was performed on vaccinated subjects with available data.
  * Pain, redness, swelling and fever were assessed in all age cohorts.
  * Drowsiness, irritability and loss of appetite were assessed in the 6 months to < 5 years cohort only.
  * Arthralgia, fatigue, headache, muscle aches and shivering were assessed in the 5 to < 18 years cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 2039 | 1149
Participants
  Pain [Any] | 1072 | 526
  Pain [Grade 3] | 31 | 19
  Redness [Any] | 421 | 233
  Redness [> 50 mm] | 16 | 4
  Swelling [Any] | 308 | 152
  Swelling [> 50 mm] | 22 | 4
  Drowsiness [Any]: number analyzed (Participants) | 691 | 697
  Drowsiness [Any] | 160 | 177
  Drowsiness [Grade 3]: number analyzed (Participants) | 691 | 697
  Drowsiness [Grade 3] | 15 | 16
  Drowsiness [Related]: number analyzed (Participants) | 691 | 697
  Drowsiness [Related] | 127 | 125
  Fever [≥37.5°C]: number analyzed (Participants) | 2039 | 1148
  Fever [≥37.5°C] | 152 | 85
  Fever [> 39°C]: number analyzed (Participants) | 2039 | 1148
  Fever [> 39°C] | 20 | 12
  Fever [Related]: number analyzed (Participants) | 2039 | 1148
  Fever [Related] | 69 | 48
  Irritability [Any]: number analyzed (Participants) | 691 | 697
  Irritability [Any] | 232 | 246
  Irritability [Grade 3]: number analyzed (Participants) | 691 | 697
  Irritability [Grade 3] | 20 | 18
  Irritability [Related]: number analyzed (Participants) | 691 | 697
  Irritability [Related] | 201 | 199
  Loss of appetite [Any]: number analyzed (Participants) | 691 | 697
  Loss of appetite [Any] | 131 | 128
  Loss of appetite [Grade 3]: number analyzed (Participants) | 691 | 697
  Loss of appetite [Grade 3] | 9 | 13
  Loss of appetite [Related]: number analyzed (Participants) | 691 | 697
  Loss of appetite [Related] | 103 | 96
  Arthralgia [Any]: number analyzed (Participants) | 1348 | 451
  Arthralgia [Any] | 85 | 30
  Arthralgia [Grade 3]: number analyzed (Participants) | 1348 | 451
  Arthralgia [Grade 3] | 2 | 1
  Arthralgia [Related]: number analyzed (Participants) | 1348 | 451
  Arthralgia [Related] | 74 | 27
  Fatigue [Any]: number analyzed (Participants) | 1348 | 451
  Fatigue [Any] | 285 | 88
  Fatigue [Grade 3]: number analyzed (Participants) | 1348 | 451
  Fatigue [Grade 3] | 15 | 6
  Fatigue [Related]: number analyzed (Participants) | 1348 | 451
  Fatigue [Related] | 225 | 72
  Headache [Any]: number analyzed (Participants) | 1348 | 451
  Headache [Any] | 218 | 76
  Headache [Grade 3]: number analyzed (Participants) | 1348 | 451
  Headache [Grade 3] | 8 | 4
  Headache [Related]: number analyzed (Participants) | 1348 | 451
  Headache [Related] | 171 | 61
  Muscle aches [Any]: number analyzed (Participants) | 1348 | 451
  Muscle aches [Any] | 410 | 133
  Muscle aches [Grade 3]: number analyzed (Participants) | 1348 | 451
  Muscle aches [Grade 3] | 6 | 3
  Muscle aches [Related]: number analyzed (Participants) | 1348 | 451
  Muscle aches [Related] | 367 | 121
  Shivering [Any]: number analyzed (Participants) | 1348 | 451
  Shivering [Any] | 45 | 17
  Shivering [Grade 3]: number analyzed (Participants) | 1348 | 451
  Shivering [Grade 3] | 2 | 1
  Shivering [Related]: number analyzed (Participants) | 1348 | 451
  Shivering [Related] | 37 | 14

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  Any = at least one symptom irrespective of intensity and relationship to vaccination; Grade 3 = preventing normal activity; Related = considered by the investigator to be causally related to the study vaccination.
Time Frame: Within 28 days following vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 2115 | 1210
Participants
  Any | 700 | 458
  Grade 3 | 102 | 62
  Related | 112 | 75

8. Secondary Outcome: Number of Subjects Reporting New Onset Chronic Illnesses and/or Serious Adverse Events (SAE)
Description: SAE: any untoward medical occurrence that
  * resulted in death,
  * was life-threatening,
  * required hospitalization or prolongation of existing hospitalization,
  * resulted in disability/incapacity, or
  * was a congenital anomaly/birth defect in the offspring of a study subject.
  Examples of possible new onset chronic illnesses include but are not limited to diabetes, asthma, allergies, autoimmune disease, cancer, neuropathic disorders.
Time Frame: Up to 6 months after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Group | Fluzone Group
Number analyzed (Participants) | 2115 | 1210
Participants
  New onset chronic illnesses | 11 | 3
  Serious adverse events | 11 | 11

ADVERSE EVENTS:
Arm/Group | Fluarix Group | Fluzone Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 11 | 11
Other Adverse Events (participants affected / at risk) | 1480/2115 | 781/1210
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Fluarix Group | Fluzone Group
Lymphadenitis (Blood and lymphatic system disorders) | 2/2115 | 0/1210
Faecaloma (Gastrointestinal disorders) | 1/2115 | 0/1210
Appendicitis (Infections and infestations) | 1/2115 | 0/1210
Cellulitis (Infections and infestations) | 1/2115 | 1/1210
Gastroenteritis (Infections and infestations) | 0/2115 | 1/1210
Gastroenteritis viral (Infections and infestations) | 0/2115 | 1/1210
Infectious mononucleosis (Infections and infestations) | 1/2115 | 0/1210
Lobar pneumonia (Infections and infestations) | 1/2115 | 0/1210
Meningitis enteroviral (Infections and infestations) | 0/2115 | 1/1210
Pharyngitis streptococcal (Infections and infestations) | 0/2115 | 1/1210
Pneumonia (Infections and infestations) | 1/2115 | 2/1210
Pneumonia viral (Infections and infestations) | 1/2115 | 0/1210
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1/2115 | 0/1210
Salmonellosis (Infections and infestations) | 1/2115 | 0/1210
Traumatic brain injury (Injury, poisoning and procedural complications) | 1/2115 | 0/1210
Dehydration (Metabolism and nutrition disorders) | 0/2115 | 1/1210
Febrile convulsion (Nervous system disorders) | 1/2115 | 2/1210
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/2115 | 0/1210
Suicide attempt (Psychiatric disorders) | 0/2115 | 1/1210
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/2115 | 0/1210
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0/2115 | 1/1210
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/2115 | 1/1210
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Group (N=2115) | Fluzone Group (N=1210)
Pyrexia (General disorders) | 102 | 86
Upper respiratory tract infection (Infections and infestations) | 116 | 74
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 81
Pain at the injection site (General disorders) | 1072 | 526
Redness at the injection site (General disorders) | 421 | 233
Swelling at the injection site (General disorders) | 308 | 152
Drowsiness (General disorders) | 160 | 177
Axillary fever (General disorders) | 152 | 85
Irritability (General disorders) | 232 | 246
Loss of appetite (General disorders) | 131 | 128
Arthralgia (General disorders) | 85 | 30
Fatigue (General disorders) | 285 | 88
Headache (General disorders) | 218 | 76
Muscle aches (General disorders) | 410 | 133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.